CLINICAL TRIAL: NCT03275623
Title: Management of Sub-Clinical Bacteriuria in Pregnancy: A Feasibility Trial
Brief Title: Management of Sub-Clinical Bacteriuria in Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Akwugo Adanna Eziefule, Staff Physician, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-17-0294
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Cystitis; Cystitis;Puerperium; Pyelonephritis
MeSH Terms: conditions — Cystitis; Pyelonephritis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic treatment (Active Comparator): Standard prenatal care with treatment for any urine culture with growth of 1- 100,000 CFU of any organism.
  Interventions: Drug: Antibiotic; Other: Standard Prenatal Care
- No antibiotic treatment (Active Comparator): Standard prenatal care without treatment for any urine culture with growth of 1- 100,000 CFU of any organism.
  Interventions: Other: Standard Prenatal Care

INTERVENTIONS:
Drug: Antibiotic — Those randomized for treatment will be prescribed the most commonly used antibiotic for urinary tract infections in pregnancy. This includes: Nitrofurantoin, Cephalexin, and Amoxicillin. It is unsure which antibiotic the participant will receive but a majority of the time it will be one of the above named antibiotic. The choice will be determined by the physician, but will accommodate participants' prior medication history and adverse events.
  Arms: Antibiotic treatment
Other: Standard Prenatal Care — Continued surveillance of urinary cultures

SUMMARY:
The purpose of the study is to determine if treatment of pregnant women with urine cultures with a low level of bacteria (less than 100,000 colony forming units (CFU)) may decrease adverse pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who seek prenatal care within the University of Texas Health System with UT Physicians.
* Urine culture of less than 100,000 CFU

Exclusion Criteria:

* Less than 18 years of age
* Risk factors to complicated UTI (including but not limited to: diverticula, urolithiasis, renal cysts, indwelling catheter, intermittent catheterization, stent placements, nephrostomy tubes, neurogenic bladder, cystocele, vesicoureteral reflux, ileal conduit)
* Use of immunosuppressant drugs
* Abnormalities of the urinary tract (including but not limited to: known ureteric or urethral strictures, tumors of the urinary tract, pelvicalyceal obstruction, congenital anomalies, history of urological procedures)
* History of renal disease including renal failure and transplants
* Urine culture > 100,000 CFU of any organism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akwugo A Eziefule, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antibiotic Treatment | No Antibiotic Treatment
Started | 30 | 30
Completed | 25 | 28
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Antibiotic Treatment | Antibiotic Treatment | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Count of Participants; unit: Participants]
  <20 | 6 | 11 | 17
  20-34 | 19 | 12 | 31
  >=35 | 5 | 7 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 17 | 15 | 32
  Hispanic | 4 | 9 | 13
  White | 5 | 4 | 9
  Other | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Have Cystitis
Description: Cystitis is defined as a urine culture with >100,000 CFU at any point during antenatal care.
Time Frame: about 10 months
Population: 2 participants in the "no antibiotic treatment" arm and 5 in the "antibiotic treatment" arm were not assessed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | No Antibiotic Treatment | Antibiotic Treatment
Number analyzed (Participants) | 28 | 25
Participants | 4 | 4

2. Primary Outcome: Number of Participants Who Have Pyelonephritis
Description: Pyelonephritis is defined as a urine culture with >100,000 CFU with fever at any point during antenatal care.
Time Frame: about 10 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | No Antibiotic Treatment | Antibiotic Treatment
Number analyzed (Participants) | 28 | 25
Participants | 3 | 4

ADVERSE EVENTS:
Time Frame: during antenatal care (about 10 months)
Arm/Group | No Antibiotic Treatment | Antibiotic Treatment
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03275623/Prot_SAP_000.pdf